CLINICAL TRIAL: NCT02602431
Title: A Unique Application of Low Laser Therapy After Third Molar Surgery: A Randomized Controlled Clinical Trial
Brief Title: Low Laser Light Therapy After Impacted Third Molar Removal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Maria Cristina Zindel Deboni, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 31861414.4.0000.0075
Record Dates: First submitted 2015-11-08; First posted 2015-11-11 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Trismus; Edema; Pain
Keywords: laser; third molar; low laser; inflammatory response
MeSH Terms: conditions — Trismus; Edema; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Extra-oral laser irradiation (Active Comparator): infra-red wave laser, 660nm, 100mW, and 107J/cm2
  Interventions: Device: Extra-oral laser irradiation
- Extra-oral placebo (Placebo Comparator): Laser point will be placed in region without irradiation on.
  Interventions: Device: Extra-oral placebo
- Intra-oral laser irradiation (Active Comparator): red wave laser, 660nm, 100mW, and 107J/cm2
  Interventions: Device: Intra-oral laser irradiation
- intra-oral placebo (Placebo Comparator): Laser point will be placed in region without irradiation on.
  Interventions: Device: Intra-oral Placebo

INTERVENTIONS:
Device: Extra-oral laser irradiation — Irradiation will be employed extra oral by infra-red wave laser, 660nm, 100mW, and 107J/cm2 in four points of Masseter muscle for 30 seconds in each
  Other Names: DMC Photon Laser III
  Arms: Extra-oral laser irradiation
Device: Intra-oral laser irradiation — Irradiation will be employed intra oral by red wave laser, 660nm, 100mW, and 107J/cm2 in four points for 30 seconds in each : 1. Superficial face of dental socket, 2. Lingual face; 3. buccal face and 4. Retromolar region
  Other Names: DMC Photn Laser III
  Arms: Intra-oral laser irradiation
Device: Extra-oral placebo — Laser point will be placed over the same extra-oral points for 30 seconds in each point without irradiation on
  Other Names: DMC Photn Laser III
  Arms: Extra-oral placebo
Device: Intra-oral Placebo — Laser point will be placed over the same intra-oral points for 30 seconds in each point without irradiation on
  Other Names: DMC Photn Laser III
  Arms: intra-oral placebo

SUMMARY:
Third molars extraction is a surgery frequently performed in dentistry. It is generally associated to a great postoperative distress rendered by pain, swelling and trismus, caused by surgical trauma inflammation. Several methods have been proposed to prevent these complications and to increase tissue repair quality. The use of low level laser therapy (LLLT) has been reported in dentistry since 1970. A large number of studies have reported the benefits of LLLT without collateral damage, positive effect as an anti-inflammatory agent and benefits in accelerating wound repair. However, some clinical applications strategies have been contradictories in everyday practice with results not always equivalent.

Objective: To verify if a single LLLT intra or extra oral application, singly, are analogous in their effects in controlling postoperative edema, trismus, pain and wound repair in third molar surgery.

DETAILED DESCRIPTION:
30 healthy participants of both genders, with 18 to 35 years-of-age, with the necessity of inferior bilateral third molar removal will be selected. Inclusion criteria will consider the presence of upper central incisive and same surgical difficulty for third molar extraction. Participants that present chronic TMJ pain, neurological or psychiatric disorders, pericoronitis, anti-inflammatory or analgesic use for the last 15 days, bisphosphonates usage history at any time, tabagism, pregnancy or a family history of photosensitivity and hypersensibility to analgesics, anti-inflammatory or antibiotics will not be included. The surgical procedures will be randomized for the group to be assigned respecting the interval of one month between the surgeries.

Intra-oral group (IO) will be that in whose participant will receive the LLLT (Photon Lase III DMC equipment) with 660 nm wavelength, 100 mW of power, 107J / cm2 of power density, during 30 seconds, positioning the tip of the laser device in straight contact with each of the four points in the surgical area:

1. corresponding to the occlusal surface of the tooth surgically extracted,
2. in the middle third of the lingual surface, point
3. the middle third of the buccal surface and point
4. retro molar triangle region. Each point will receive energy 3J (Et= 12J).

The extra-oral group (EO) will receive phototherapy with the 808nm of wavelength following the same above protocol although positioning the laser point over the skin in straight contact with four points on the masseter muscle:

1. next jaw insert,
2. lower middle region,
3. upper middle region
4. near the insertion of the zygomatic arch.

In the IO group the extra-oral region will not be irradiated (the laser tip will be put in place without energy) in the EO group it will be done the opposite, so as the same patient will be the control because the participant will not be capable to identify which group he belongs to. The same investigator will perform surgical procedures and laser therapy. All participants will receive the same postoperative medication. Three distances will evaluate the range of edema: from tragus to the corner of the mouth, from gonial angle to the corner of the mouth and from gonial angle to the corner of the eye using a malleable millimeter rule. Trismus will be evaluated by the maximum range of mouth opening considering the inter-incisal distance between the edges of upper and lower right central incisors by a caliper in three moments: before surgery, 24 hours and 8 days after surgery. Participants will be asked to fill in a diary to assess the severity of postoperative pain on a visual analogue pain scale after the end of anesthetic effect: 4, 6, 8, 24, 48 hours postoperatively. The amount and time of medication will be also recorded. The quality of wound repair will be evaluated by two blinded calibrated observers, 24 hours and 8 days postoperatively in score from 0 to 3. The data will be submitted to appropriate statistical analysis for non-parametric samples.

ELIGIBILITY:
Inclusion Criteria:

* necessity of bilateral impacted third molar removal with similar dental arch positioning and similar surgical difficulty.

Exclusion Criteria:

* Compromised Systemic Health status, Neurologic and/or mental disorders, local infection history, anti-inflammatory or analgesic use for the last 15 days, tabagism, ethylism, pregnancy.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Scores on the Visual Analog scale | 4, 6, 8, 24, 48hours post operative period
  measurements in a diary after anesthetic sensation had stopped and 4, 6, 8, 24, 48hours post operatively

SECONDARY OUTCOMES:
Edema percentage | 24 hours after surgery
  measurement of face parameters dimension pre and post operative
mouth aperture in millimeters | 24 hours after surgery
  comparison between maximum mouth aperture pre and post operatively

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cristina Deboni, PhD, Principal Investigator — Associate Professor
Locations (1):
- Maria Cristina Zindel Deboni, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Larrazabal C, Garcia B, Penarrocha M, Penarrocha M. Influence of oral hygiene and smoking on pain and swelling after surgical extraction of impacted mandibular third molars. J Oral Maxillofac Surg. 2010 Jan;68(1):43-6. doi: 10.1016/j.joms.2009.07.061. PMID 20006153
- [Background] Mehrabi M, Allen JM, Roser SM. Therapeutic agents in perioperative third molar surgical procedures. Oral Maxillofac Surg Clin North Am. 2007 Feb;19(1):69-84, vi. doi: 10.1016/j.coms.2006.11.010. PMID 18088865
- [Background] Markovic A, Todorovic Lj. Effectiveness of dexamethasone and low-power laser in minimizing oedema after third molar surgery: a clinical trial. Int J Oral Maxillofac Surg. 2007 Mar;36(3):226-9. doi: 10.1016/j.ijom.2006.10.006. Epub 2006 Dec 8. PMID 17157479
- [Background] Aras MH, Gungormus M. Placebo-controlled randomized clinical trial of the effect two different low-level laser therapies (LLLT)--intraoral and extraoral--on trismus and facial swelling following surgical extraction of the lower third molar. Lasers Med Sci. 2010 Sep;25(5):641-5. doi: 10.1007/s10103-009-0684-1. Epub 2009 May 31. PMID 19484402
- [Background] Brignardello-Petersen R, Carrasco-Labra A, Araya I, Yanine N, Beyene J, Shah PS. Is adjuvant laser therapy effective for preventing pain, swelling, and trismus after surgical removal of impacted mandibular third molars? A systematic review and meta-analysis. J Oral Maxillofac Surg. 2012 Aug;70(8):1789-801. doi: 10.1016/j.joms.2012.01.008. Epub 2012 Mar 6. PMID 22398186
- [Background] He WL, Yu FY, Li CJ, Pan J, Zhuang R, Duan PJ. A systematic review and meta-analysis on the efficacy of low-level laser therapy in the management of complication after mandibular third molar surgery. Lasers Med Sci. 2015 Aug;30(6):1779-88. doi: 10.1007/s10103-014-1634-0. Epub 2014 Aug 7. PMID 25098769
- [Background] Kazancioglu HO, Ezirganli S, Demirtas N. Comparison of the influence of ozone and laser therapies on pain, swelling, and trismus following impacted third-molar surgery. Lasers Med Sci. 2014 Jul;29(4):1313-9. doi: 10.1007/s10103-013-1300-y. Epub 2013 Mar 14. PMID 23494104
- [Background] Lopez-Ramirez M, Vilchez-Perez MA, Gargallo-Albiol J, Arnabat-Dominguez J, Gay-Escoda C. Efficacy of low-level laser therapy in the management of pain, facial swelling, and postoperative trismus after a lower third molar extraction. A preliminary study. Lasers Med Sci. 2012 May;27(3):559-66. doi: 10.1007/s10103-011-0936-8. Epub 2011 May 27. PMID 21617973
- [Background] Ferrante M, Petrini M, Trentini P, Perfetti G, Spoto G. Effect of low-level laser therapy after extraction of impacted lower third molars. Lasers Med Sci. 2013 May;28(3):845-9. doi: 10.1007/s10103-012-1174-4. Epub 2012 Jul 28. PMID 22843310
- [Background] Pallotta RC, Bjordal JM, Frigo L, Leal Junior EC, Teixeira S, Marcos RL, Ramos L, Messias Fde M, Lopes-Martins RA. Infrared (810-nm) low-level laser therapy on rat experimental knee inflammation. Lasers Med Sci. 2012 Jan;27(1):71-8. doi: 10.1007/s10103-011-0906-1. Epub 2011 Apr 12. PMID 21484455